CLINICAL TRIAL: NCT06841926
Title: A Study to Evaluate the Pharmacokinetics of ZX-7101A for Suspension Versus Tablets in a Single Oral Administration Under Fasting Conditions in Healthy Chinese Adult Male Subjects
Brief Title: Study to Evaluate the Pharmacokinetics and Relative Bioavailability of Metabolites in Healthy Chinese Adult Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Nanjing Zenshine Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ZX-7101A-213
Record Dates: First submitted 2025-02-13; First posted 2025-02-24 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Respiratory Viral Infection

STUDY DESIGN:
Intervention Model Description: The study was a single-center, randomized, open-label, two-dose, two-cycle, two-sequence, double-crossover design.
  A total of 40 healthy male subjects were randomly divided into 2 sequences, 20 subjects in each sequence. Subjects received 40 mg of test preparation ZX-7101A dry suspension (4 bags) or 40 mg of reference preparation ZX-7101A tablets (1 tablet) per cycle.
  Subjects received either the test formulation (T) or the reference formulation (R) orally in the first cycle according to their random allocation of subjects, and crossed over to the reference formulation (R) or the test formulation (T) in the second cycle. The cleaning period was at least 21 days between the two weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The test preparation was followed by the reference preparation (Other): Group 1: The test preparation was followed by the reference preparation:
  20 subjects were given the test formulation (T) : ZX-7101A dry suspension 40 mg (4 bags) orally in the first cycle, and crossed over to the reference formulation ZX-7101A tablets 40 mg (1 tablet) in the second cycle, with a wash period of at least 21 days between two weeks.
  Interventions: Drug: ZX-7101A dry suspension; Other: ZX-7101A tablet
- The reference preparation was followed by the test preparation (Other): Group 2: The reference preparation was followed by the test preparation:
  20 subjects were given reference formulation ZX-7101A tablets 40 mg (1 tablet) orally in the first cycle, and crossed over to the the test formulation (T) : ZX-7101A dry suspension 40 mg (4 bags) in the second cycle, with a wash period of at least 21 days between two weeks.
  Interventions: Drug: ZX-7101A dry suspension; Other: ZX-7101A tablet

INTERVENTIONS:
Drug: ZX-7101A dry suspension — Test formulation (T) : ZX-7101A dry suspension Specification: 10 mg/ bag Dosage：40 mg (4 bags)、 once
Other: ZX-7101A tablet — Reference formulation (R): ZX-7101A tablet Specification: 40 mg/ tablet Dosage：40 mg (1 tablet)、 once

SUMMARY:
Study to evaluate the pharmacokinetics and relative bioavailability of metabolites in healthy Chinese adult males

DETAILED DESCRIPTION:
To evaluate the pharmacokinetic profile and relative bioavailability of the active metabolite ZX-7101 (parent drug) after a single oral administration of 40 mg ZX-7101A for suspension and 40 mg ZX-7101A tablet in healthy Chinese adult male subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects aged 18 to 45 years (including the cut-off value, subject to the signing of the informed consent)
* Body mass index (BMI) of 19 to 26 kg/m2 (including the cut-off value), with a body weight of at least 50 kg
* Based on the medical history, physical examination, vital signs, 12-lead electrocardiogram, laboratory tests (blood routine, urine routine, blood biochemistry, coagulation function), viral serology and chest X-ray results, the investigator judged that the subjects were in good general health (normal or abnormal examination results were not clinically significant).
* Voluntary informed consent, no fertility and sperm donation plans within 90 days after the last dose of medication, and voluntary use of highly effective contraception (including a partner) (Nonpharmacologic contraception was required during the clinical trial)
* Before signing the informed consent, the patients should have a full understanding of the trial content, process and possible adverse reactions, and voluntarily sign the informed consent.
* Be able to complete the study in accordance with the protocol requirements

Exclusion Criteria:

* Allergic (multiple drug and food allergies) or those who are likely to be allergic to the investigational drug or any component of the investigational drug as judged by the investigator;
* Subjects with taste and smell dysfunction
* Oral ulcer or mucosal injury
* Subjects with a previous or present medical history of clinically abnormal metabolic, hepatic, renal, hematologic, pulmonary, cardiovascular, gastrointestinal, urinary, endocrine, neurologic, or psychiatric disease who were deemed by the investigator to be ineligible for participation in the study
* Subjects whose vital signs were abnormal and clinically significant before administration
* Subjects with abnormal white blood cell or neutrophil count before administration that was judged by the investigators to be clinically significant;
* Before administration, the subjects had abnormal liver function: total bilirubin >1.5× upper limit of normal (ULN), AST >1.5× ULN, ALT >1.5× ULN;
* Estimated glomerular filtration rate <90 mL/min/1.73 m2 (eGFR formula)
* QTc interval > 450ms (Fridericia's correction, QTcF=QT/(RR^0.33)), QRS>120ms
* Acute respiratory infection within 2 weeks before the study
* Subjects who have difficulty swallowing drugs or have a history of gastrointestinal diseases that seriously affect drug absorption (including but not limited to reflux esophagitis, chronic diarrhea, inflammatory bowel disease, etc.); Or have a history of gastrointestinal surgery or resection that may alter the absorption and/or excretion of oral medications (subjects who have undergone appendectomy may be included)
* Use of any prescription drug or Chinese herbal medicine within 4 weeks before trial initiation and use of over-the-counter or nutrual products (including multivalent cations, inhibitors, and metal supplements) within 2 weeks before trial initiation would require a longer interval of at least 5 half-ages of the drug
* Subjects who had consumed more than 14 units of alcohol per week (1 unit =360 mL of beer or 45 mL of 40% spirits or 150 mL of wine) in the 6 months before screening or had received a positive breath test for alcohol
* Smoking more than five cigarettes per day or habitual use of nicotine-containing products in the 3 months before screening.
* Subjects who were unwilling to abstain from foods or drinks containing caffeine or alcohol that affect drug metabolism within 72 hours before drug administration and during the period of observation in phase I ward.
* Use of any known liver enzyme inducer or liver enzyme inhibitor (grapefruit, orange juice, etc.) within 14 days before administration.
* Subjects with a history of drug abuse (morphine, dimethyldioxyamphetamine, methamphetamines, tetrahydrocannabinol, ketamine, cocaine) or screening positive for drug abuse;
* Subjects who were serologically positive for syphilis antibody (TP-trust), hepatitis B surface antigen, hepatitis C virus antibody or human immunodeficiency virus antibody;
* Donating >400 mL within 3 months or >200 mL within 4 weeks prior to the screening period or planning to donate during the study period;
* Those who have difficulty in venous blood collection;
* Subjects who participated in other clinical trials or used any other clinical trial drugs or devices within 3 months before screening;
* Vaccinated within 1 month prior to dose or planned to be vaccinated during the study period;
* Subjects who had a surgical procedure within 6 months before screening or who were scheduled to undergo surgery during the trial;
* Any other situation that the investigator considers may affect the subject's provision of informed consent or compliance with the trial protocol or completion of the trial according to the study process, or the subject's participation in the trial may affect the trial results or their own safety.Subjects who were serologically positive for syphilis antibody (TP-trust), hepatitis B surface antigen, hepatitis C virus antibody or human immunodeficiency virus antibody;

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-02-20 (Actual); Primary Completion 2025-04-18 (Actual); Study Completion 2025-04-18 (Actual)

PRIMARY OUTCOMES:
The pharmacokinetic parameters Cmax of the active metabolite ZX-7101 (parent drug) | From Day1 up to Day 36
  Pharmacokinetic parameters Cmax of the active metabolite ZX-7101 (parent drug) in plasma after administration of ZX-7101A dry suspension /ZX-7101A tablets
The pharmacokinetic parameters AUC0-t of the active metabolite ZX-7101 (parent drug) | From Day1 up to Day 36
  Pharmacokinetic parameters AUC0-t of the active metabolite ZX-7101 (parent drug) in plasma after administration of ZX-7101A dry suspension /ZX-7101A tablets
The pharmacokinetic parameters AUC0-inf of the active metabolite ZX-7101 (parent drug) | From Day1 up to Day 36
  Pharmacokinetic parameters AUC0-inf of the active metabolite ZX-7101 (parent drug) in plasma after administration of ZX-7101A dry suspension /ZX-7101A tablets
Relative bioavailability of the active metabolite ZX-7101 (parent drug) | From Day1 up to Day 36
  Relative bioavailability of the active metabolite ZX-7101 (parent drug) in plasma after administration of ZX-7101A dry suspension /ZX-7101A tablets.

SECONDARY OUTCOMES:
Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v5.0 | From Day 1 up to Day 36
  To evaluate the safety and tolerability of a single oral administration of ZX-7101A dry suspension (40 mg/tablet) in healthy Chinese adult male subjects
Cmax | From Day 1 up to Day 36
  To evaluate the pharmacokinetic: Cmax of ZX-7101A (prodrug) after a single oral administration of ZX-7101A dry suspension 40 mg and ZX-7101A tablets 40 mg in healthy Chinese adult male subjects
AUC0-t | From Day 1 up to Day 36
  To evaluate the pharmacokinetic: AUC0-t of ZX-7101A (prodrug) after a single oral administration of ZX-7101A dry suspension 40 mg and ZX-7101A tablets 40 mg in healthy Chinese adult male subjects
AUC0-inf | From Day 1 up to Day 36
  To evaluate the pharmacokinetic:AUC0-inf of ZX-7101A (prodrug) after a single oral administration of ZX-7101A dry suspension 40 mg and ZX-7101A tablets 40 mg in healthy Chinese adult male subjects
Evaluation of palatability | On Day 1
  The proportion of all subjects who received ZX-7101A dry suspension with a score ≥50 (including not good not bad, good, very good)
Tmax | From Day 1 up to Day 36
  PK parameters of prodrug ZX-7101A and its active metabolite ZX-7101 (parent drug) : Tmax
Vz/F | From Day 1 up to Day 36
  PK parameters of prodrug ZX-7101A and its active metabolite ZX-7101 (parent drug) : Vz/F
CL/F | From Day 1 up to Day 36
  PK parameters of prodrug ZX-7101A and its active metabolite ZX-7101 (parent drug) : CL/F
t1/2 | From Day 1 up to Day 36
  PK parameters of prodrug ZX-7101A and its active metabolite ZX-7101 (parent drug) : t1/2
λz | From Day 1 up to Day 36
  PK parameters of prodrug ZX-7101A and its active metabolite ZX-7101 (parent drug) : λz

CONTACTS AND LOCATIONS:
Locations (1):
- West China Second University Hospital, Sichuan University and Children's Hospital Zhejiang University School of Medicine, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No